CLINICAL TRIAL: NCT03093038
Title: Early Stability of the Delta-TT Cup With Polyethylene Insert Compared to the Delta-TT Cup With Ceramic Insert. A Randomised RSA Study
Brief Title: Early Stability of the Delta-TT Cup With Polyethylene Insert Versus a Ceramic Insert. A RSA Study.
Acronym: RSA-DELTA-TT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JointResearch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL44230.100.13 - v1.0
Record Dates: First submitted 2014-12-17; First posted 2017-03-28 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- H-MAX stem & Delta-TT cup + polyethylene (Active Comparator): H-MAX femoral stem and the Delta-TT cup with polyethylene insert
  Interventions: Device: H-MAX stem & Delta-TT cup + polyethylene
- H-MAX stem & Delta-TT cup + ceramic (Experimental): H-MAX femoral stem and the Delta-TT cup with ceramic insert
  Interventions: Device: H-MAX stem & Delta-TT cup + ceramic
- C2 stem & Delta-TT cup + ceramic (Experimental): C2 femoral stem and the Delta-TT cup with ceramic insert
  Interventions: Device: C2 stem & Delta-TT cup + ceramic

INTERVENTIONS:
Device: H-MAX stem & Delta-TT cup + polyethylene — H-MAX femoral stem & Delta-TT cup with a polyethylene insert
  Arms: H-MAX stem & Delta-TT cup + polyethylene
Device: H-MAX stem & Delta-TT cup + ceramic — H-MAX femoral stem & Delta Delta-TT cup with a Ceramic insert
  Arms: H-MAX stem & Delta-TT cup + ceramic
Device: C2 stem & Delta-TT cup + ceramic — C2 femoral stem Delta Delta-TT cup with a Ceramic insert
  Arms: C2 stem & Delta-TT cup + ceramic

SUMMARY:
The goal of this study is to study the stability of the Delta-TT cup with polyethylene insert and the Delta-TT cup with ceramic insert both combined with the H-MAX femoral stem by means of RSA to assess whether the differences in stiffness of the cup will have an influence on incorporation and mechanical stability.

It is hypothesized that there will be more micromotion on the short-term (<2 years) in the patients with the ceramic insert because of the higher stiffness, however, all components will be considered stable on the short and long-term.

DETAILED DESCRIPTION:
Rationale: Roentgen Stereophotogrammetric Analysis (RSA) is a very accurate measurement technique used to obtain micromotion of the implants relative to inserted tantalum markers in the surrounding bone. Using RSA, long-term predictions of prosthetic loosening can be made based on a two years follow-up. Therefore, it is recommended to analyse all (new) prosthetic components by means of RSA.

Objective: The goal of this study is to study in a randomised trial the stability of the Delta-TT cup with polyethylene insert and the Delta-TT cup with ceramic insert both combined with the H-MAX femoral stem by means of RSA to assess whether the differences in stiffness of the cup will have an influence on incorporation and mechanical stability. It is hypothesized that there will be more micromotion on the short-term (<2 years) in the patients with the ceramic insert because of the higher stiffness, however, all components will be considered stable on the short and long-term. Secondary goal is to compare the stability of the C2 femoral stem, to the H-MAX femoral stem as well as to compare it to relevant migration results of similar stems from the literature. These RSA results will contribute to knowledge about the early stability and long-term prosthetic loosening of these cementless stems.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo primary total hip replacement.
* Patient is able to understand the meaning of the study and is willing to sign the ethical committee approved, study-specific Informed Patient Consent Form.
* Ability and willingness to follow instructions and to return for follow-up evaluations.
* The subject is a male or non-pregnant female between 18 and 75 years of age.

Exclusion Criteria:

* The subject is morbidly obese, defined as Body Mass Index (BMI) of > 40.
* The subject will be operated bilaterally.
* Patients having a deformity or disease located in other joints than the hip that needs surgery and is limiting their ability to walk.
* The subject has an active or suspected latent infection in or about the hip joint.
* The subject has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* The subject has a systemic or metabolic disorder leading to progressive bone deterioration.
* The subject's bone stock is compromised by disease or infection which cannot provide adequate support and/or fixation to the prosthesis.
* Female patients planning a pregnancy during the course of the study.
* The patient is unable or unwilling to sign the Informed Consent specific to this study.
* Subject deemed unsuitable for participation in the study based on the investigator's judgement.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in stability | 2 years
  Stability will be assessed with Roentgen Stereophotogrammetric Analysis (RSA). RSA will be used to determine the micromotion of the femur and cup components with respect to the bone.The RSA data of the components will be described in terms of translational and rotational movements.

SECONDARY OUTCOMES:
Change from Baseline in Quality of Life | 2 years
  Quality of Life (QoL) will be assessed with the questionaire EuroQoL 5D (EQ- 5D)
Change from Baseline in Quality of Life | 5 years
  Quality of Life (QoL) will be assessed with the questionaire EuroQoL 5D (EQ- 5D)
Change from Baseline in Physical Function | 2 years
  Physical Function will be assessed with the Hip disability and Osteoarthritis Outcome Score - Physical Function Short Form (HOOS-PS)
Change from Baseline in Physical Function | 5 years
  Physical Function will be assessed with the Hip disability and Osteoarthritis Outcome Score - Physical Function Short Form (HOOS-PS)
Change from Baseline in Physical Function and Pain | 2 years
  Physical Function will be assessed with the Oxford Hip Score (OHS)
Change from Baseline in Physical Function and Pain | 5 years
  Physical Function will be assessed with the Oxford Hip Score (OHS)
Change from Baseline in Pain | 2 years
  Pain will be assessed with a Numeric Rating Scale (NRS)
Change from Baseline in Pain | 5 years
  Pain will be assessed with a Numeric Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf W Poolman, MD PhD, Principal Investigator — Onze Lieve Vrouwe Gasthuis
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klaassen AD, van Loon J, Willigenburg NW, Koster LA, Kaptein BL, van der Hulst VPM, Haverkamp D, Moojen DJF, Poolman RW. Comparison of 5-year cup and stem migration between ceramic-on-ceramic and ceramic-on-polyethylene bearing in press-fit total hip arthroplasty: a randomised controlled trial using radiostereometric analysis. Hip Int. 2024 Nov;34(6):701-716. doi: 10.1177/11207000241265653. Epub 2024 Aug 19. PMID 39160668